CLINICAL TRIAL: NCT04406649
Title: An Open-Label, 12-Month Study to Evaluate the Safety and Tolerability of STS101 (Dihydroergotamine Nasal Powder) in the Acute Treatment of Migraine
Brief Title: A Study to Evaluate the Safety of STS101 in the Acute Treatment of Migraine
Acronym: ASCEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Satsuma Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS101-003
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura
Keywords: dihydroergotamine; dihydroergotamine mesylate; migraine
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STS101 (Experimental): STS101 (dihydroergotamine nasal powder)
  Interventions: Drug: Dihydroergotamine

INTERVENTIONS:
Drug: Dihydroergotamine — Dihydroergotamine is a semi-synthetic derivative of ergotamine tartrate.
  Other Names: Dihydroergotamine Mesylate

SUMMARY:
Study STS101-003 is a multi-center, multiple dose (PRN), open-label, 12-month study to evaluate the safety and tolerability of STS101 (dihydroergotamine nasal powder) in the acute treatment of migraine.

DETAILED DESCRIPTION:
The ASCEND trial is a multi-center, multiple dose (PRN), open-label, 12-month study to evaluate the safety and tolerability of STS101 (dihydroergotamine nasal powder) in the acute treatment of migraine.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, 18-65 years of age at the time of Screening Visit
* Subject has at least 1-year history of migraines (with or without aura), according to the
* International Classification of Headache Disorder, 3rd Edition (ICHD3)

Key Exclusion Criteria:

* Pregnant or breast-feeding women
* Women of child-bearing potential not using or not willing to use highly effective contraception.
* Diagnosis of headache conditions other than migraine with or without aura, including diagnosis of basilar or hemiplegic migraines or cluster headache.
* History of coronary artery disease, coronary artery vasospasm (including Printz-metals' angina), clinically significant arrhythmia or, peripheral vascular disease, ischemic disease (e.g. Raynaud's syndrome, ischemic bowel syndrome, angina pectoris, myocardial infarction, or documented silent ischemia); percutaneous coronary intervention, or cardiac surgery.
* History of cerebrovascular disease, including but not limited to stroke, transient ischemic attack, cerebral hemorrhage, subarachnoid hemorrhage.
* Diagnosis of major depression with current symptoms, psychosis, alcohol abuse or dependence, drug abuse or dependence, major psychiatric conditions (e.g. schizophrenia, psychosis or Bipolar disorder), dementia. Other significant neurological or psychiatric disorders (including other pain syndromes or risk of suicide) that in the opinion of the investigator might interfere with study participation and assessments or subject safety.
* Any clinically significant symptoms or conditions, including but not limited to central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator might interfere with study assessments or safety of participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Albrecht, MD, Study Chair — Satsuma Pharmaceuticals, Inc.
Locations (44):
- United States (44):
  - WR-PRI, Encino, California
  - Collaborative Neuroscience, Long Beach, California
  - WR-PRI, Los Alamitos, California
  - Downtown LA Research, Los Angeles, California
  - Clinical Research Institute, Los Angeles, California
  - WR-PRI, Newport Beach, California
  - Hillcrest Medical Research, DeLand, Florida
  - MD Clinical, Hallandale, Florida
  - Multi-Specialty Research Associates, Lake City, Florida
  - ClinCloud, Maitland, Florida
  - Biotech Pharmaceuticals, Miami, Florida
  - Behavioral Clinical Research, Miami Lakes, Florida
  - CNS Health Care - Orlando, Orlando, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Infinity Clinical Research, Sunrise, Florida
  - Santos Research Center, Corp, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Clinical Research CF, Winter Haven, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Integrated Clinical Trial Services, Inc, West Des Moines, Iowa
  - Delricht Research, Prairieville, Louisiana
  - Medvadis Research at Boston PainCare Center, Waltham, Massachusetts
  - Healthcare Research Network, Hazelwood, Missouri
  - Clinvest Research, Springfield, Missouri
  - Montana Medical Research, Missoula, Montana
  - Wake Research - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Neurology Headache Clinic, Lebanon, New Hampshire
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - SPRI Clinical Research, Brooklyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Neurology Diagnosis, Dayton, Ohio
  - Delricht Research, Tulsa, Oklahoma
  - Thomas Jefferson University/Jefferson Headache Center, Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - CNS Healthcare - Memphis, Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - DM Clinical Research, Tomball, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Georgetown University Hospital, Department of Neurology, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tepper SJ, Albrecht D, Ailani J, Kirby L, Strom S, Rapoport AM. Long-Term (12-Month) Safety and Tolerability of STS101 (Dihydroergotamine Nasal Powder) in the Acute Treatment of Migraine: Data from the Phase 3 Open-Label ASCEND Study. CNS Drugs. 2024 Dec;38(12):1017-1027. doi: 10.1007/s40263-024-01118-8. Epub 2024 Oct 7. PMID 39373843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 54 sites in the United States.
Pre-assignment Details: A total of 482 participants were enrolled in the study (all enrolled subjects population).
Groups:
- STS101 5.2 mg: Subjects received a single oral dose of STS101 (dihydroergotamine nasal powder) 5.2 mg.
Period: Overall Study
Arm/Group | STS101 5.2 mg
Started | 482
Completed | 205
Not Completed | 277

BASELINE CHARACTERISTICS:
Population: The data are from All Subjects (Mk1/Mk2 device) Safety Population.
Arm/Group | STS101 5.2 mg
Number analyzed (Participants) | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 389
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 47
  White | 379
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 446

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Attacks With Sustained Freedom From Headache Pain 2-48 Hours (Modified Intent to Treat Population)
Description: The subject's rating was documented on a four-point scale from no pain (= 0), mild pain (= 1), moderate pain (= 2) to severe pain (= 3). Pain freedom means the pain went from moderate (2) or severe (3) to no pain (0).
Time Frame: At Month 12 of Study Medication Dosing
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 5.2 mg
Number analyzed (Participants) | 183
Participants | 40.0

2. Primary Outcome: Percentage of Participants With Attacks With Sustained Freedom From Most Bothersome Symptom 2-48 Hours (Modified Intent to Treat Population)
Description: Subjects were prompted to document the presence of 3 symptoms (photophobia, phonophobia, and nausea) immediately before study drug administration and during the treated migraine attack.
Time Frame: At Month 12 of Study Drug Administration
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 5.2 mg
Number analyzed (Participants) | 183
Participants | 60

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year.
Description: The all subjects (Mk1/Mk2 device) safety population was used for adverse event reporting.
Arm/Group | STS101 5.2 mg
All-Cause Mortality (participants affected / at risk) | 0/446
Serious Adverse Events (participants affected / at risk) | 3/446
Other Adverse Events (participants affected / at risk) | 206/446
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STS101 5.2 mg (N=446)
Acute Myocardial infarction (Cardiac disorders) | 1
Postural Orthostatic Tachycardia Syndrome (Cardiac disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | STS101 5.2 mg (N=446)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 64
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 30
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23
COVID-19 (Infections and infestations) | 25
Dysgeusia (Nervous system disorders) | 33
Nausea (Gastrointestinal disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT04406649/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04406649/SAP_001.pdf